CLINICAL TRIAL: NCT05176470
Title: A Phase IB Study to Assess the Safety and Efficacy of Neoadjuvant Administration of Autologous Tumor Infiltrating Lymphocytes (LN144/Lifileucel) and Pembrolizumab for Treatment of Patients With Locally Advanced (Stage IIIB-D)/Metastatic (Stage IV) Melanoma
Brief Title: Neoadj Admin Autologous Tumor Infiltrating Lymphocytes & Pembrolizumab for Treatment of Adv Melanoma Patients
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Richard Wu (Other)
Collaborators: Iovance Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Richard Wu, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-21202; NCI-2021-11063 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-12-17; First posted 2022-01-04 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Locally Advanced Melanoma; Pathologic Stage IIIB Cutaneous Melanoma AJCC v8; Pathologic Stage IIIC Cutaneous Melanoma AJCC v8; Pathologic Stage IIID Cutaneous Melanoma AJCC v8; Stage IV Melanoma
Keywords: Adoptive T-cell Therapy; Melanoma; Neoadjuvant; Tumor-infiltrating Lymphocytes; LN-144; Lifileucel
MeSH Terms: conditions — Melanoma | interventions — Cyclophosphamide; fludarabine; lifileucel; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab, lifileucel) (Experimental): Patients receive pembrolizumab IV on day -14, cyclophosphamide IV QD on days -7 to -6, fludarabine IV over 30 minutes QD on days -5 to -1, and lifileucel IV infusion on day 0. Patients also receive pembrolizumab IV on day 28 and 70, and undergo surgery on day 80.
  MAINTENANCE: Patients receive pembrolizumab IV every 6 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Lifileucel; Biological: Pembrolizumab; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Biological: Lifileucel — Given by IV infusion
  Other Names: Autologous TIL LN-144; Autologous Tumor Infiltrating Lymphocytes LN-144; Contego; LN-144
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This phase I/II trial tests the safety and side effects of LN-144 (Lifileucel) and pembrolizumab in treating patients with stage IIIB-D or stage IV melanoma that has spread to nearby tissue or lymph nodes. Biological therapies, such as LN-144 (Lifileucel), use substances made from living organisms that may attack specific tumor cells and stop them from growing or kill them. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving lifileucel and pembrolizumab may make the tumor smaller.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of the neoadjuvant administration of Pembrolizumab and LN-144 (Lifileucel) isolated from tumor-involved metastatic lymph node(s) in 3 stage IIIB-D melanoma patients. (Part 1) II. To evaluate the safety profile and surgical tolerability of MK-3475 (pembrolizumab) and LN-144 (Lifileucel) in 12 patients, as measured by the incidence of grade >= 3 treatment-emergent adverse events (TEAEs). (Part 2)

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of Pembrolizumab and LN-144(Lifileucel) in 12 patients by determining the overall objective response rate (ORR), using the Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) and immune-related RECIST (irRECIST) criteria, as assessed by the investigator. (Part 2 only) II. To further evaluate the efficacy of Pembrolizumab and LN-144 (Lifileucel) in 12 patients using the 24-month relapse-free survival rate (RFS), using RECIST 1.1 and irRECIST, as assessed by the investigator. (Part 2 only)

EXPLORATORY OBJECTIVES:

I. To determine rates of major pathologic response (MPR) for high-risk stage IIIB-D melanoma patients treated with neoadjuvant administration of MK-3475 (pembrolizumab) and LN-144 (Lifileucel).

II. To determine the association between the proportion of PD-1+CD4+ or CD8+ tumor infiltrating lymphocytes (TILs) isolated from tumor involved lymph node(s) via flow cytometry, and probability of MPR, ORR, and RFS.

III. To determine the association between neoantigen specificity and probability of MPR, ORR, and RFS.

IV. To determine the correlation between tumor mutation burden (TMB) and MPR, ORR, and RFS.

V. To determine the correlation between intratumoral IFN-gamma and T-effector gene signatures and probability of MPR, ORR, and RFS.

VI. To evaluate the correlation between serum cytokines (IL-8, IL-6), and probability of MPR, ORR, and RFS.

VII. To evaluate the success rates of growing TILs from lymph node metastases, and the potential predictive factors (i.e., patient's age, CD8/CD4 ratios, inhibitory receptor expressions).

VIII. To correlate the doses of TILs infused to patients and the probability of MPR, ORR, and RFS.

IX. To perform additional translational studies utilizing the unstained slides or FFPE (paraffin blocks) on the resected melanoma tumor specimen post LN-144 (Lifileucel) neoadjuvant therapy.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) on day -14, cyclophosphamide IV once daily (QD) on days -7 to -6, fludarabine IV over 30 minutes QD on days -5 to -1, and lifileucel IV infusion on day 0. Patients also receive pembrolizumab IV on day 28 and 70, and undergo surgery on day 80.

MAINTENANCE: Patients receive pembrolizumab IV every 6 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 to 75 years of age
* Must have a confirmed diagnosis of Stage IIIB-D locally advanced or Stage IV melanoma (American Joint Committee on Cancer [AJCC] 8th edition) with measurable disease in the lymph node(s) documented by computed tomography (CT) or ultrasound imaging (>= 15 mm short axis) or by physical exam. Patients must also have measurable primary site of disease, including cutaneous and/or intransit metastases by imRECIST (>= 20 mm chest x-ray [CXR], >= 10 mm CT, or >= 10 mm by exam)
* No prior therapy is allowed
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 and an estimated life expectancy of >= 3 months in the opinion of the investigator
* Patients must have at least one easily accessible measurable tumor-involved lymph node(s) documented by CT or ultrasound imaging for TIL harvest
* Patients must be amenable to have ultrasound examination of measurable lymph node(s) and have pathologic confirmation of melanoma metastases in the lymph node (fine needle aspiration [FNA] acceptable) in the 28 days preceding the first administration of the treatment
* Patients with and without BRAF V600E/K mutations are included.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
* Patients with a history of herpes simplex virus (HSV) infection must have been treated. Patients with a history of Epstein-Barr virus (EBV) or cytomegalovirus (CMV) infection must be asymptomatic and have low viral loads
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional classification. To be eligible for this trial, patients should be class 2B or better
* Women must not be pregnant or breast-feeding due to potential harm to an unborn fetus and possible risk of adverse events in nursing infants with the anti-PD-1 regimen(s) being used.

  * All females of childbearing potential must have a blood test or urine study within 14 days prior to registration to rule out pregnancy.
  * A female of childbearing potential is defined as any woman, regardless of sexual orientation, or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy, or 3) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding consecutive months)
* Women of childbearing potential and sexually active males must not conceive or father children by using accepted and effective method(s) of contraception or by abstaining from sexual intercourse from the time of study registration and continuing until at least 5 months after the last dose of anti-PD-1 treatment for female patients and for at least 7 months after the last dose of anti-PD-1 treatment for male patients who are sexually active with a woman of childbearing potential (WOCBP).
* Patients must have adequate organ and marrow function as defined below at study enrollment and prior to surgical resection. (these labs must be obtained ≤ 4 weeks prior to protocol registration and ≤1 week prior to surgery):
* Hemoglobin >= 10 g/dL
* Neutrophils >= 1500/ul
* Leukocytes >= 3000/ul
* Lymphocytes >= 700/ul
* Blood platelet >= 100,000/ul
* Serum creatinine =< 1.5 x upper limit of normal or creatinine clearance (CrCl) >= 40 mL/min (if using the Cockcroft-Gault formula)
* Serum bilirubin =< 2.0 mg/dL
* Total bilirubin =< 1.5 x upper limit of normal (except for patients with Gilbert syndrome, who can have total bilirubin < 3 mg/dL)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2 x upper limit of normal
* Lactate dehydrogenase (LDH) =< 1.5 x upper limit of normal
* Patients (or legally authorized representative) must have the ability to understand the requirements of the study, have provided written informed consent as evidenced by signature on an informed consent form (ICF) approved by an Institutional Review Board/Independent Ethics Committee (IRB/IEC), and agree to abide by the study restrictions and return to the site for the required assessments, including the RFS Follow-up Period

Exclusion Criteria:

* Ocular/uveal melanoma
* Chemotherapy or radiotherapy within 4 weeks before baseline (6 weeks for nitroso-urea and mitomycin C)
* Contraindication for the use of vasopressor agents
* Patients with HIV active infection or seropositivity are excluded. Patients with active Hep B or Hep C based on serology and viral load are excluded. Patients with active CMV or EBV based on serology and viral load are excluded.
* History or current manifestation of severe progressive heart disease (congestive heart failure with LVEF < 50% by echocardiogram or MUGA scan, coronary artery disease, uncontrolled arterial hypertension, uncontrolled arrhythmia, or myocardial infarction in the past 6 months.
* Patients with active interstitial lung disease (ILD)/pneumonitis or a history of ILD/pneumonitis requiring treatment with systemic steroids.
* Patients should be excluded if they had prior treatment with an anti- PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways.
* Patients who have a history of hypersensitivity to immune checkpoint therapy drug(s) or any component or excipient of LN-144 or other study drugs:

  * Nivolumab, pembrolizumab, or related products
  * Any monoclonal antibody
  * NMA-LD preconditioning regimen (cyclophosphamide, mesna, and fludarabine)
  * Proleukin, aldesleukin, IL-2
  * Antibiotics (ABX) of the aminoglycoside group (i.e., streptomycin, gentamicin); except those who are skin-test negative for gentamicin hypersensitivity
  * Any component of the LN-144 infusion product formulation including dimethyl sulfoxide (DMSO), human serum albumin (HSA), IL-2, and dextran-40
* History of chronic autoimmune disease (Addison's disease, multiple sclerosis, Graves' disease, rheumatoid arthritis, systemic lupus erythematosus, etc…) except patient with active vitiligo or a history of vitiligo. Patients with history of psoriasis is allowed
* History of inflammatory bowel disease, celiac disease, or other chronic gastrointestinal conditions associated with diarrhea.
* Patients who have had another primary malignancy within the previous 3 years (except for those which do not require treatment or have been curatively treated >1 year ago, and in the judgment of the Investigator, does not pose a significant risk of recurrence including, but not limited to, non-melanoma skin cancer, DCIS, LCIS, prostate cancer Gleason score ≤6).
* Any serious, acute or chronic illness (i.e., active infection) needing antibiotics administration, coagulation's disorders, or any medical disorder requiring unauthorized concomitant treatment described in this study.
* Positive serology for HTLV1/HTLV2, or syphilis.
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days before study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if > 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (eg, contrast dye allergy) or for treatment of non-autoimmune conditions (eg, delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
* Patients who have obstructive or restrictive pulmonary disease and have a documented forced expiratory volume in 1 second (FEV1) of ≤ 60% of predicted normal:

  * If a patient is not able to perform reliable spirometry due to abnormal upper airway anatomy (i.e., tracheostomy), a 6- minute walk test may be used to assess pulmonary function.
  * Patients who are unable to walk a distance of at least 80% predicted for age and sex or demonstrates evidence of hypoxia at any point during the test (SpO2 < 90%) are excluded.
* Active infections, including COVID-19, within 30 days, unless deemed fully resolved/treated by the study PI.
* Participated in another clinical study with an investigational product within 21 days of the initiation of treatment.
* Adults under a legal protection regime (i.e., guardianship, trusteeship).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of neoadjuvant administration of MK-3475 and LN-144/Lifileucel in 3 stage IIIB-D melanoma patients (Phase 1) | Up to 2 years
  Success rate of tumor infiltrating lymphocyte (TIL) expansion from all screened eligible patients who have had tumor-involved lymph node(s) removed; percentage of all eligible patients who have completed the screening and treated with LN-144/lifileucel.
Incidence of grade >= 3 treatment-emergent adverse events (both immune and non-immune related) (Phase 2) | Up to 2 years
  The severity of AEs will be graded according to CTCAE version 5.0, and frequencies and percentages of patients with AEs will be tabulated by severity grade.

SECONDARY OUTCOMES:
Overall objective response rate | Up to 2 years
  Evaluated by Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) and immune-related RECIST (irRECIST) criteria.
Relapse-free survival (RFS) rate | At 24 months
  Kaplan-Meier method will be used to estimate the median time and the corresponding 95% CI.

OTHER OUTCOMES:
Major pathologic response (MPR) rate | Up to 2 years
  MPR will be summarized by number and percentage of patients with major pathologic response, as well as the corresponding 2-sided exact 95% confidence intervals (95% CI).
Immune correlates (as described above) with respect to response and 24-month relapse free survival, of the TIL/LN-144 + pembrolizumab neoadjuvant therapy | Up to 2 years
Success rate of TIL growth from tumor-involved lymph node(s) | Up to 2 years
Doses of the infused TIL with respect to response and 24-month relapse-free survival | Up to 2 years
Changes in the patients' health-related quality of life | Up to 2 years
  Measured by a standardized questionnaire during and after the study protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Wu, M.D. Ph.D., Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (1):
  • Informed Consent Form (2023-10-16): https://cdn.clinicaltrials.gov/large-docs/70/NCT05176470/ICF_000.pdf